CLINICAL TRIAL: NCT01558882
Title: Impact of Essure Tubal Sterilization Devices on the Endometrium
Status: Terminated | Type: Observational
Why Stopped: Trouble with recruting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/VL-05; 2012-A00253-40 (Other: RCB number)
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Sterilization, Tubal
Keywords: Essure; Change in uterine cytokines; Change in uterine natural killer cells; cytokine; natural killer cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All left over samples will be included in the hematology biological collection at the Nîmes University Hospital.
  Endometrial flushing samples will also be included in the Nîmes University Hospital biobank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 10 patients: The patients included desire tubal sterilization via the ESSURE technique.
  Interventions: Device: Essure

INTERVENTIONS:
Device: Essure — Essure devices are deployed according to manufacturer's instructions for tubal sterilization.

SUMMARY:
The mobilization of natural killer cells (uNK) triggers and coordinates all stages of embryo implantation. They are at the origin of the local secretion of cytokines, growth factors, chemokines affecting vascular development and the local immunotrophisme for the conceptus. The main objective of this study is to evaluate the expression of endometrial uNK cells before and after tubal obstruction by Essure devices. Endoluminal and endometrial levels of various cytokines and growth factors will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow up
* The patient has had at least one child
* The patient desires definitive tubal sterilization via the ESSURE technique
* The legal delay of 4 months between request for sterilization and surgery has been respected
* Local contraception (condom or spermicide) must be used for three months before and after tubal sterilization

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient had a diagnosed pregnancy (this includes pregnancies lost or interruptions in the 2nd or 3rd trimester) within the 4 months before ESSURE implants
* The patient has a contraindication for a treatment used in this study
* The patient uses one of the following types of contraception: intrauterine device; oestroprogestatif (pill).
* Endometriosis
* Gynecological infection
* adenomyosis
* uterine polyp
* uterine surgery

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten women desiring tubal sterilization via the ESSURE method.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2014-11-28 (Actual); Study Completion 2014-11-28 (Actual)

PRIMARY OUTCOMES:
Change in number of uNK/CD56 cells per field | baseline (Day 0) - 3 months
  Number of cells per field from endometrial biopsy

SECONDARY OUTCOMES:
% change in IL-1 beta titration in uterine flushing sample | baseline (day 0) - 3 months
% change in IL-12 titration in uterine flushing sample | baseline (day 0) - 3 months
% change in IL-15 titration in uterine flushing sample | baseline (day 0) - 3 months
% change in IL-18 titration in uterine flushing sample | baseline (day 0) - 3 months
% change in TWEAK titration in uterine flushing sample | baseline (day 0) - 3 months
% change in TNF-alpha titration in uterine flushing sample | baseline (day 0) - 3 months
% change in G-CSF titration in uterine flushing sample | baseline (day 0) - 3 months
% change in G-CSF receptor titration in uterine flushing sample | baseline (day 0) - 3 months
% change in VEGF titration in uterine flushing sample | baseline (day 0) - 3 months
Change in the number of macrophage cells per field on endometrial biopsy | baseline (day 0) to 3 months
Change in the number of T cells per field on endometrial biopsy | baseline (day 0) to 3 months
Change in expression of IL-1 beta in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of IL-12 in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of IL-15 in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of IL-18 in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of TWEAK in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of TNF-alpha in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of G-CSF in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of G-CSF receptor in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of VEGF in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of beta-2 microglobulin in endometrial biopsy | baseline (day 0) to 3 months
Change in expression of RPL13A (reference gene) in endometrial biopsy | baseline (day 0) to 3 months
Change in endometrial volume (cm^3) | baseline (day 0) to 3 months
Change in subendometrial vascular flow index | baseline (day 0) to 3 months
Time needed for Essure deployment (minutes) | baseline (day 0), immediatly after intervention
Type of anesthesia used for Essure deployment | baseline (day 0), immediatly after intervention
Number of spirals visible in the left uterine cavity after Essure deployment | baseline (day 0), immediatly after intervention
Number of spirals visible in the right uterine cavity after Essure deployment | baseline (day 0), immediatly after intervention
Presence/absence of bilateral tube obstruction | 3 months
Change in number of uNK/CD56 cells per field | 2 months before intervention - Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - APHP - Hôpital Antoine Beclere, Clamart
  - APHP - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes